CLINICAL TRIAL: NCT03280381
Title: Randomized Crossover Trial of the Nifty Feeding Cup and a Medicine Cup in Preterm Infants Who Have Difficulty Breastfeeding
Brief Title: Nifty Feeding Cup Versus Generic Medicine Cup Preterm Infants Who Have Difficulty Breastfeeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Seattle Children's Hospital (Other); Komfo Anokye Teaching Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 978912-3
Record Dates: First submitted 2017-09-06; First posted 2017-09-12 (Actual); Results first posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Infant,Premature; Feeding; Difficult, Newborn
Keywords: Nifty Cup; breastfeeding difficulties; preterm infant; cup feeding
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Investigators will conduct a randomized crossover trial in mothers/caregivers with a preterm infant in the mother-baby unit at Komfo Anokye Teaching Hospital (KATH) in Kumasi, Ghana. Each caregiver/infant pair will use the Nifty Feeding Cup for two feeds and the standardized generic cup for two feeds. Cross-over means each caregiver/infant pair will use both cups, with the order of the cup used first and second randomized.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NIFTY Feeding Cup First (Experimental): Each caregiver/infant pair will first use the Nifty Feeding Cup for two feeds and then the standardized generic cup for two feeds.
  Interventions: Other: Nifty feeding cup; Other: Generic medicine cup
- Generic Medicine Cup First (Experimental): Each caregiver/infant pair will first use the standardized generic cup for two feeds and then the Nifty Feeding Cup for two feeds.
  Interventions: Other: Nifty feeding cup; Other: Generic medicine cup

INTERVENTIONS:
Other: Nifty feeding cup — The 40 mL Nifty Feeding Cup features an extended reservoir off the lip of the cup that holds a small bolus of milk, ensuring efficient delivery of milk, is made of a durable, soft, silicone material that protects the infant's mouth from injury, has embossed measurements help with tracking volume and intake of milk, is ergonomically designed for frequent use and to enhance finger and wrist control of milk flow and is made from a quick-drying, ultraviolet radiation-resistant, durable, affordable silicone that can be boiled for sterilization. Mothers can directly express into the cup, reducing possible cross-contamination from other containers.
Other: Generic medicine cup — The generic cup that will be used in this study is a small medicine cup 30 ml in size.Small medicine cups are manufactured by a variety of manufacturers and are commonly used in health facilities to feed breastmilk to infants who are having breastfeeding difficulties. The cups are generally translucent, calibrated with a variety of measurements including 2.5-30 mL.

SUMMARY:
The investigators will establish an evidence base for the Nifty Feeding Cup by evaluating its effectiveness and caregiver satisfaction. The investigators will conduct a randomized crossover trial that compares the Nifty Feeding Cup to a standardized, generic medicine cup used to feed preterm infants with breastfeeding difficulties at Komfo Anokye Teaching Hospital (KATH) in Kumasi, Ghana.

DETAILED DESCRIPTION:
The investigators aim to compare the Nifty Feeding Cup to a standardized, generic cup in up to 200 preterm infants. The aim and hypotheses were selected based on the most informative outcomes given the scope of the funding. The investigators will test the hypotheses that Nifty Feeding Cup feeding compared to generic cup feeding will result in:

1. Less spillage
2. Greater caregiver satisfaction
3. Shorter duration of feeds

ELIGIBILITY:
Inclusion Criteria:

Infant

* Born preterm (<37 weeks gestational age) at time of birth
* Corrected gestational age is <37 weeks per the modified Dubowitz score on date of enrollment
* Diagnosed with feeding difficulties
* Patient in the mother-baby unit at KATH
* Clinically indicated to start cup feeding (including an infant who has a nasogastric tube and is cup feeding or indicated to start cup feeding)
* Has an anticipated hospital stay that is at least 48 hours

Caregiver:

* At least 18 years of age
* One of the following biologic family members of the infant (Mother, Grandmother, Aunt)
* Self-identifies as the primary feeder of the infant
* Prior experience feeding the potential infant participant with nipple feeding (e.g. breast feeding, bottle feeding) or nasogastric [NG] tube
* Verifies willingness to comply with all study procedures

Exclusion Criteria:

Infant

* Congenital anomaly except for minor anomalies (e.g. an extra digit or ear tag is okay)
* Other condition or situation that makes infant unlikely to be able to comply with study procedures. Examples include the infant anticipated to not be in hospital long enough, infant has a suspected intestinal obstruction, or necrotizing enterocolitis.
* No mother, grandmother, or aunt caregiver available to participate in study
* Enrolled in another study at KATH that would interfere with his/her ability to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2018-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christy McKinney, Ph.D., Principal Investigator — Seattle Children's Hospital
Locations (1):
- Komfo Anokye Teaching Hospital (KATH), Kumasi, Ghana

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- NIFTY Feeding Cup First: Each caregiver/infant pair will first use the Nifty Feeding Cup for two feeds and then the standardized generic cup for two feeds.
  Nifty Feeding Cup: The 40 mL cup features an extended reservoir off the lip of the cup that holds a small bolus of milk, has embossed measurements to track volume and intake of milk, is ergonomically designed for frequent use and to enhance finger and wrist control of milk flow and is made from a quick-drying, ultraviolet radiation-resistant, durable, affordable and soft silicone that can be boiled for sterilization. Mothers can directly express into the cup, reducing possible cross-contamination from other containers.
  Generic medicine cup: A generic 30 mL small medicine cup was used in this study. Small medicine cups are manufactured by many manufacturers and are generally translucent and calibrated with a variety of measurements. They are commonly used in health facilities to feed breastmilk to infants who are having breastfeeding difficulties.
- Generic Medicine Cup First: Each caregiver/infant pair will first use the standardized generic cup for two feeds and then the Nifty Feeding Cup for two feeds.
  Nifty Feeding Cup: The 40 mL cup features an extended reservoir off the lip of the cup that holds a small bolus of milk, has embossed measurements to track volume and intake of milk, is ergonomically designed for frequent use and to enhance finger and wrist control of milk flow and is made from a quick-drying, ultraviolet radiation-resistant, durable, affordable and soft silicone that can be boiled for sterilization. Mothers can directly express into the cup, reducing possible cross-contamination from other containers.
  Generic medicine cup: A generic 30 mL small medicine cup was used in this study. Small medicine cups are manufactured by many manufacturers and are generally translucent and calibrated with a variety of measurements. They are commonly used in health facilities to feed breastmilk to infants who are having breastfeeding difficulties.
Period: Overall Study
Arm/Group | NIFTY Feeding Cup First | Generic Medicine Cup First
Started | 101 | 99
Completed | 101 | 97
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Generic Medicine Cup First: Each caregiver/infant pair will first use the Nifty Feeding Cup for two feeds and then the standardized generic cup for two feeds.
  Nifty Feeding Cup: The 40 mL cup features an extended reservoir off the lip of the cup that holds a small bolus of milk, has embossed measurements to track volume and intake of milk, is ergonomically designed for frequent use and to enhance finger and wrist control of milk flow and is made from a quick-drying, ultraviolet radiation-resistant, durable, affordable and soft silicone that can be boiled for sterilization. Mothers can directly express into the cup, reducing possible cross-contamination from other containers.
  Generic medicine cup: A generic 30 mL small medicine cup was used in this study. Small medicine cups are manufactured by many manufacturers and are generally translucent and calibrated with a variety of measurements. They are commonly used in health facilities to feed breastmilk to infants who are having breastfeeding difficulties.
- Total: Total of all reporting groups
Arm/Group | NIFTY Feeding Cup First | Generic Medicine Cup First | Total
Number analyzed (Participants) | 101 | 99 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 101 | 99 | 200
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline demographic data
  Participants
    Female | 101 | 99 | 200
    Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Caregiver Satisfaction [Immediate]
Description: Caregiver's satisfaction will be the cup she prefers, which will be recorded in the In-Hospital Preference Survey completed after the caregiver has finished the feeding portion of the study. Data refers to number of caregivers who prefer the Nifty Cup.
Time Frame: 24-36 hours
Measure: Number; unit: participants
Arm/Group | NIFTY Feeding Cup First | Generic Medicine Cup First
Number analyzed (Participants) | 101 | 97
participants | 82 | 67

2. Primary Outcome: Spillage
Description: Spillage will be reported as a percent with the amount of milk in grams spilled/mopped up divided by the total amount of milk weighed in grams less the total amount of milk not used. Each caregiver-infant pair will be provided with a bib cloth for each observed feeding. The bib cloth will be weighed before and after each feed and the weights recorded on the Feeding Assessment form. The difference between the pre and post weights will be used as the measure of the amount spilled. A digital scale will be used to measure the milk weight, which will be recorded in grams.
Time Frame: 24-36 hours
Measure: Mean (Standard Deviation); unit: percentage of feed spilled
Arm/Group | NIFTY Feeding Cup First | Generic Medicine Cup First
Number analyzed (Participants) | 101 | 97
percentage of feed spilled | 8.9 (6.9) | 9.3 (8.7)

ADVERSE EVENTS:
Time Frame: Data were collected over the time it took mothers to feed their infants twice with each cup, an average of 13 minutes per feed.
Arm/Group | NIFTY Feeding Cup First | Generic Medicine Cup First
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/99
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/99
Other Adverse Events (participants affected / at risk) | 0/101 | 0/99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-24): https://cdn.clinicaltrials.gov/large-docs/81/NCT03280381/Prot_SAP_000.pdf